CLINICAL TRIAL: NCT00758264
Title: Immunogenicity & Safety Study of GSK Biologicals' Meningococcal Vaccine GSK134612 When Co-administered With GSK Biologicals' Pneumococcal Vaccine GSK1024850A in Healthy 12-23-month-old Children Previously Primed With GSK1024850A
Brief Title: Co-administration of Meningococcal Vaccine GSK134612 and Pneumococcal Vaccine GSK1024850A vs Individual Administration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111393
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2018-05-09 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2017-04

CONDITIONS: Infections, Meningococcal
Keywords: Safety; Routine infancy vaccination; Meningococcal vaccine; Immunogenicity; Pneumococcal vaccine
MeSH Terms: conditions — Meningococcal Infections

ARMS (3):
- Group A (Experimental): Meningococcal vaccine GSK134612 co-administered with pneumococcal vaccine GSK1024850A.
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Pneumococcal vaccine GSK1024850A
- Group B (Active Comparator): Pneumococcal vaccine GSK1024850A followed one month later by meningococcal vaccine GSK134612.
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Pneumococcal vaccine GSK1024850A
- Group C (Active Comparator): Meningococcal vaccine GSK134612 followed one month later by pneumococcal vaccine GSK1024850A.
  Interventions: Biological: Meningococcal vaccine GSK134612; Biological: Pneumococcal vaccine GSK1024850A

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 — Single dose intramuscular injection.
Biological: Pneumococcal vaccine GSK1024850A — Single dose intramuscular injection.

SUMMARY:
The purpose of this study is to demonstrate, in 12-23 months old subjects, the non-inferiority of meningococcal vaccine GSK134612 and pneumococcal vaccine GSK1024850A when co-administered, compared to each vaccine administered individually.

DETAILED DESCRIPTION:
Multi-center study with 3 parallel groups. One group will receive 2 vaccines injections at the same visit (pneumococcal+ meningococcal), one group will receive a pneumococcal vaccine followed one month later by a meningococcal vaccine, and the last group will receive the meningococcal vaccine followed one month later by the pneumococcal vaccine.

All subjects will have one blood sample taken before vaccination and one blood sample taken one month after each vaccination (i.e. the first group will have 2 blood samples taken, and the other two groups will have 3 blood sample taken)

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female between, and including, 12 and 23 months of age at the time of the first booster vaccination, who previously participated in study 109661 conducted in Mexico or in study 109861 conducted in Taiwan and who received 3 doses of the GSK1024850A vaccine.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine(s), or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days before the first dose of vaccine(s) and 30 days after the last dose of vaccine(s).
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Previous vaccination with a meningococcal vaccine.
* Previous administration of a fourth dose of a pneumococcal vaccine
* Previous vaccination with tetanus toxoid within the last month (including also tetanus toxoid given as part of Hib-TT conjugate vaccine).
* History of meningococcal or pneumococcal invasive disease.
* History of reactions or allergic disease likely to be exacerbated by any component of the vaccines.
* Hypersensitivity reaction due to previous vaccination with GSK1024850A vaccine.
* History of seizures (this criterion does not apply to subjects who have had a single, uncomplicated febrile convulsion in the past) or progressive neurological disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection, based on medical history and physical examination (no laboratory testing required).
* A family history of congenital or hereditary immunodeficiency, unless the child has previously been documented, through laboratory testing, to have normal immune function.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 363 (Actual)
Dates: Start 2008-10-30; Primary Completion 2009-06-02 (Actual); Study Completion 2009-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Mexico (2):
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
- Taiwan (2):
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan Hsien

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Huang LM et al. Immunogenicity and safety of PHiD-CV coadministered with a candidate meningococcal tetanus toxoid conjugate vaccine (MenACWY-TT) in children previously primed with PHiD. Abstract presented at the 5th Asian Congress of Pediatric Infectious Diseases (ACPID). Taipei, Taiwan, 23-26 September 2010.
- [Background] Ruiz-Palacios GM, Huang LM, Lin TY, Hernandez L, Guerrero ML, Villalobos AL, Van der Wielen M, Moreira M, Fissette L, Borys D, Miller JM. Immunogenicity and safety of a booster dose of the 10-valent pneumococcal Haemophilus influenzae protein D conjugate vaccine coadministered with the tetravalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine in toddlers: a randomized trial. Pediatr Infect Dis J. 2013 Jan;32(1):62-71. doi: 10.1097/INF.0b013e3182784143. PMID 23076383
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 111393 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111393 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111393 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111393 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111393 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111393 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111393 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 subjects have not been contacted for the Extended Safety Follow Up phase, out of which 2 subjects have not been contacted due to lost to follow-up (1 subject in Nimenrix + Synflorix Group and 1 subject in Nimenrix Group) and 1 subject due to consent withdrawal (Synflorix Group).
Groups:
- Nimenrix + Synflorix Group: Subjects aged 12 to 23 months, male or female, primed with Synflorix vaccine who received Nimenrix vaccine and Synflorix booster vaccine at Month 0. Both vaccines were administered intramuscularly, in the right thigh for the Nimenrix conjugate vaccine, in the left thigh for the Synflorix vaccine.
- Nimenrix Group: Subjects aged 12 to 23 months, male or female, primed with Synflorix vaccine who received Nimenrix conjugate vaccine at Month 0 and Synflorix booster vaccine at Month 1. Both vaccines were administered intramuscularly, in the right thigh for the Nimenrix conjugate vaccine, in the left thigh for the Synflorix vaccine.
- Synflorix Group: Subjects aged 12 to 23 months, male or female, primed with Synflorix vaccine who received Synflorix booster vaccine at Month 0 and Nimenrix conjugate vaccine at Month 1. Both vaccines were administered intramuscularly, in the right thigh for the Nimenrix conjugate vaccine, in the left thigh for the Synflorix vaccine.
Period: Active Phase
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Started | 182 | 91 | 90
Completed | 181 | 91 | 85
Not Completed | 1 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Other | 0 | 0 | 4
Period: Extended Safety Follow Up (ESFU) Phase
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Started | 181 | 90 | 89
Completed | 181 | 90 | 89
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group | Total
Number analyzed (Participants) | 182 | 91 | 90 | 363
Age, Continuous [Mean (Standard Deviation); unit: Months] | 17.2 (1.97) | 17.2 (1.88) | 17.4 (1.86) | 17.25 (1.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 56 | 47 | 186
  Male | 99 | 35 | 43 | 177
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 91 | 46 | 46 | 183
  Asian - East Asian heritage | 91 | 45 | 44 | 180

OUTCOME MEASURES:

1. Primary Outcome: Anti-pneumococcal Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in micrograms per milliliter (µg/mL). Anti-pneumococcal serotypes assessed were Anti-1, Anti-4, Anti-5, Anti-6B, Anti-7F, Anti-9V, Anti-14, Anti-18C, Anti-19F and Anti-23F via the 22F-inhibition Enzyme Linked Immunosorbent Assay (ELISA).
Time Frame: At Month 1
Population: The analysis was done on the According-to-protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available. The primary outcome concerns the Nimenrix + Synflorix Group and the Synflorix Group.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 175 | 81 | 81
μg/mL
  Anti-1: number analyzed (Participants) | 175 | 76 | 81
  Anti-1 | 3.43 [3.06 to 3.85] | 0.33 [0.27 to 0.41] | 3.60 [2.96 to 4.38]
  Anti-4: number analyzed (Participants) | 172 | 75 | 79
  Anti-4 | 6.86 [6.06 to 7.76] | 0.52 [0.41 to 0.65] | 6.98 [5.82 to 8.37]
  Anti-5: number analyzed (Participants) | 175 | 78 | 81
  Anti-5 | 4.97 [4.40 to 5.62] | 0.54 [0.43 to 0.67] | 5.07 [4.34 to 5.93]
  Anti-6B: number analyzed (Participants) | 175 | 76 | 80
  Anti-6B | 2.91 [2.48 to 3.41] | 0.53 [0.41 to 0.68] | 3.14 [2.55 to 3.85]
  Anti-7F: number analyzed (Participants) | 175 | 78 | 79
  Anti-7F | 5.32 [4.75 to 5.95] | 0.88 [0.74 to 1.04] | 5.10 [4.26 to 6.10]
  Anti-9V: number analyzed (Participants) | 175 | 80 | 80
  Anti-9V | 4.70 [4.15 to 5.32] | 0.79 [0.64 to 0.98] | 4.74 [3.96 to 5.67]
  Anti-14: number analyzed (Participants) | 175 | 76 | 80
  Anti-14 | 8.89 [7.65 to 10.33] | 1.16 [0.88 to 1.51] | 9.00 [7.40 to 10.95]
  Anti-18C: number analyzed (Participants) | 175 | 77 | 78
  Anti-18C | 9.81 [8.40 to 11.45] | 0.73 [0.56 to 0.94] | 19.48 [15.20 to 24.97]
  Anti-19F: number analyzed (Participants) | 175 | 78 | 80
  Anti-19F | 19.16 [16.60 to 22.12] | 1.39 [1.00 to 1.92] | 20.79 [17.67 to 24.45]
  Anti-23F: number analyzed (Participants) | 174 | 81 | 81
  Anti-23F | 4.46 [3.80 to 5.25] | 0.59 [0.43 to 0.81] | 3.79 [2.94 to 4.88]
Statistical Analysis 1: Comparison: Nimenrix + Synflorix Group vs Synflorix Group; Demonstration of non-inferiority of Synflorix vaccine when co-administered with Nimenrix conjugate vaccine versus Synflorix vaccine given alone (Nimenrix conjugate vaccine was administered 1 month later) in terms of anti-pneumococcal serotype 1 antibody concentrations; Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit (LL) of the 95% confidence interval (CI) of the geometric mean concentration (GMC) ratio between the Nimenrix +Synflorix Group and the Synflorix Group (Nimenrix + Synflorix Group over Synflorix Group) is above (>) 0.5; Adjusted GMC ratio = 0.87, 95% CI 2-sided [0.72 to 1.05]
Statistical Analysis 2: Comparison: Nimenrix + Synflorix Group vs Synflorix Group; Demonstration of non-inferiority of Synflorix vaccine when co-administered with Nimenrix conjugate vaccine versus Synflorix vaccine given alone (Nimenrix conjugate vaccine was administered 1 month later) in terms of anti-pneumococcal serotype 4 antibody concentrations; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Adjusted GMC ratio = 1.03, 95% CI 2-sided [0.84 to 1.26]
Statistical Analysis 3: Comparison: Nimenrix + Synflorix Group vs Synflorix Group; Demonstration of non-inferiority of Synflorix vaccine when co-administered with Nimenrix conjugate vaccine versus Synflorix vaccine given alone (Nimenrix conjugate vaccine was administered 1 month later) in terms of anti-pneumococcal serotype 5 antibody concentrations; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Adjusted GMC ratio = 0.90, 95% CI 2-sided [0.74 to 1.10]
Statistical Analysis 4: Comparison: Nimenrix + Synflorix Group vs Synflorix Group; Demonstration of non-inferiority of Synflorix vaccine when co-administered with Nimenrix conjugate vaccine versus Synflorix vaccine given alone (Nimenrix conjugate vaccine was administered 1 month later) in terms of anti-pneumococcal serotype 6B antibody concentrations; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Adjusted GMC ratio = 0.84, 95% CI 2-sided [0.66 to 1.07]
Statistical Analysis 5: Comparison: Nimenrix + Synflorix Group vs Synflorix Group; Demonstration of non-inferiority of Synflorix vaccine when co-administered with Nimenrix conjugate vaccine versus Synflorix vaccine given alone (Nimenrix conjugate vaccine was administered 1 month later) in terms of anti-pneumococcal serotype 7F antibody concentrations; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Adjusted GMC ratio = 1.00, 95% CI 2-sided [0.84 to 1.20]
Statistical Analysis 6: Comparison: Nimenrix + Synflorix Group vs Synflorix Group; Demonstration of non-inferiority of Synflorix vaccine when co-administered with Nimenrix conjugate vaccine versus Synflorix vaccine given alone (Nimenrix conjugate vaccine was administered 1 month later) in terms of anti-pneumococcal serotype 9V antibody concentrations; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Adjusted GMC ratio = 0.94, 95% CI 2-sided [0.78 to 1.14]
Statistical Analysis 7: Comparison: Nimenrix + Synflorix Group vs Synflorix Group; Demonstration of non-inferiority of Synflorix vaccine when co-administered with Nimenrix conjugate vaccine versus Synflorix vaccine given alone (Nimenrix conjugate vaccine was administered 1 month later) in terms of anti-pneumococcal serotype 14 antibody concentrations; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Adjusted GMC ratio = 0.98, 95% CI 2-sided [0.78 to 1.23]
Statistical Analysis 8: Comparison: Nimenrix + Synflorix Group vs Synflorix Group; Demonstration of non-inferiority of Synflorix vaccine when co-administered with Nimenrix conjugate vaccine versus Synflorix vaccine given alone (Nimenrix conjugate vaccine was administered 1 month later) in terms of anti-pneumococcal serotype 18C antibody concentrations; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Adjusted GMC ratio = 0.52, 95% CI 2-sided [0.41 to 0.67]
Statistical Analysis 9: Comparison: Nimenrix + Synflorix Group vs Synflorix Group; Demonstration of non-inferiority of Synflorix vaccine when co-administered with Nimenrix conjugate vaccine versus Synflorix vaccine given alone (Nimenrix conjugate vaccine was administered 1 month later) in terms of anti-pneumococcal serotype 19F antibody concentrations; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Adjusted GMC ratio = 0.86, 95% CI 2-sided [0.68 to 1.08]
Statistical Analysis 10: Comparison: Nimenrix + Synflorix Group vs Synflorix Group; Demonstration of non-inferiority of Synflorix vaccine when co-administered with Nimenrix conjugate vaccine versus Synflorix vaccine given alone (Nimenrix conjugate vaccine was administered 1 month later) in terms of anti-pneumococcal serotype 23F antibody concentrations; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Adjusted GMC ratio = 1.07, 95% CI 2-sided [0.83 to 1.38]

2. Primary Outcome: Number of Subjects With Serum Bactericidal Assay Using Rabbit Complement Against Neisseria Meningitides Serogroups A, C , W-135, Y (rSBA-MenA, rSBA-MenC, rSBA-MenW -135 and rSBA-Men-Y) Antibody Titers Greater Than or Equal to (≥) the Cut-off Value
Description: The cut-off value for the rSBA titers was greater than or equal to (≥) 1:8.
Time Frame: At Month 1
Population: The analysis was done on the According-to-protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available. The primary outcome concerns the Nimenrix + Synflorix Group and the Nimenrix Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 174 | 80 | 79
Participants
  rSBA-MenA: number analyzed (Participants) | 174 | 80 | 63
  rSBA-MenA | 173 | 78 | 23
  rSBA-MenC: number analyzed (Participants) | 174 | 80 | 76
  rSBA-MenC | 173 | 79 | 9
  rSBA-MenW-135: number analyzed (Participants) | 174 | 80 | 74
  rSBA-MenW-135 | 174 | 79 | 40
  rSBA-MenY | 173 | 80 | 48
Statistical Analysis 1: Comparison: Nimenrix + Synflorix Group vs Nimenrix Group; Demonstration of non-inferiority of Nimenrix conjugate vaccine when co-administered with Synflorix vaccine versus Nimenrix conjugate vaccine given alone (Synflorix vaccine was administered 1 month later) in terms of serum bactericidal assay using rabbit complement against Neisseria meningitides serogroup A (rSBA-MenA); Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit (LL) of the 2-sided standardized asymptotic 95% confidence interval (CI) for the group difference in percentage of subjects with serum bactericidal antibody using baby rabbit complement against Neisseria meningitides serogroup A (rSBA-MenA) titer ≥ 1:8 (Nimenrix + Synflorix Group minus Nimenrix Group) is ≥ -10%; Difference in percentage = 1.93, 95% CI 2-sided [-1.09 to 8.15]
Statistical Analysis 2: Comparison: Nimenrix + Synflorix Group vs Nimenrix Group; Demonstration of non-inferiority of Nimenrix conjugate vaccine when co-administered with Synflorix vaccine versus Nimenrix conjugate vaccine given alone (Synflorix vaccine was administered 1 month later) in terms of serum bactericidal assay using rabbit complement against Neisseria meningitides serogroup C (rSBA-MenC); Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit (LL) of the 2-sided standardized asymptotic 95% confidence interval (CI) for the group difference in percentage of subjects with serum bactericidal antibody using baby rabbit complement against Neisseria meningitides serogroup C (rSBA-MenC) titer ≥ 1:8 (Nimenrix + Synflorix Group minus Nimenrix Group) is ≥ -10%; Difference in percentage = 0.68, 95% CI 2-sided [-2.11 to 6.22]
Statistical Analysis 3: Comparison: Nimenrix + Synflorix Group vs Nimenrix Group; Demonstration of non-inferiority of Nimenrix conjugate vaccine when co-administered with Synflorix vaccine versus Nimenrix conjugate vaccine given alone (Synflorix vaccine was administered 1 month later) in terms of serum bactericidal assay using rabbit complement against Neisseria meningitides serogroup W-135 (rSBA-MenW-135); Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit (LL) of the 2-sided standardized asymptotic 95% confidence interval (CI) for the group difference in percentage of subjects with serum bactericidal antibody using baby rabbit complement against Neisseria meningitides serogroup W-135 (rSBA-MenW-135) titer ≥ 1:8 (Nimenrix + Synflorix Group minus Nimenrix Group) is ≥ -10%; Difference in percentage = 1.25, 95% CI 2-sided [-0.94 to 6.76]
Statistical Analysis 4: Comparison: Nimenrix + Synflorix Group vs Nimenrix Group; Demonstration of non-inferiority of Nimenrix conjugate vaccine when co-administered with Synflorix vaccine versus Nimenrix conjugate vaccine given alone (Synflorix vaccine was administered 1 month later) in terms of serum bactericidal assay using rabbit complement against Neisseria meningitides serogroup Y (rSBA-MenY); Test type: Non-Inferiority — Non-inferiority was demonstrated if the lower limit (LL) of the 2-sided standardized asymptotic 95% confidence interval (CI) for the group difference in percentage of subjects with serum bactericidal antibody using baby rabbit complement against Neisseria meningitides serogroup Y (rSBA-MenY) titer ≥ 1:8 (Nimenrix + Synflorix Group minus Nimenrix Group) is ≥ -10%; Difference in percentage = 0.00, 95% CI 2-sided [-2.18 to 4.6]

3. Primary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-Men-Y Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs) and are measured in titers.
Time Frame: At Month 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 174 | 80 | 79
Titers
  rSBA-MenA: number analyzed (Participants) | 174 | 80 | 63
  rSBA-MenA | 6673.7 [5680.7 to 7840.4] | 5016.6 [3594.8 to 7000.8] | 23.5 [12.7 to 43.5]
  rSBA-MenC: number analyzed (Participants) | 174 | 80 | 76
  rSBA-MenC | 2496.6 [2096.5 to 2973.0] | 2044.0 [1522.8 to 2743.6] | 6.4 [4.7 to 8.7]
  rSBA-MenW- 135: number analyzed (Participants) | 174 | 80 | 74
  rSBA-MenW- 135 | 11731.0 [10270.7 to 13398.9] | 8407.7 [6225.4 to 11355.0] | 35.8 [21.5 to 59.6]
  rSBA-MenY: number analyzed (Participants) | 173 | 80 | 79
  rSBA-MenY | 6797.8 [6014.4 to 7683.4] | 5606.2 [4484.5 to 7008.3] | 68.4 [39.9 to 117.2]

4. Secondary Outcome: Anti-pneumococcal Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in micrograms per milliliter (µg/mL). The pneumococcal serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Anti-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) via 22F-inhibition ELISA. GMCs post Dose 2 are not presented for Nimenrix + Synflorix Group, as they received only one study vaccination dose.
Time Frame: Before vaccination (PRE) and at one month post dose 2 (Month 2)
Population: The analysis was done on the According-to-protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 168 | 81 | 78
μg/mL
  Anti-1, PRE: number analyzed (Participants) | 167 | 76 | 76
  Anti-1, PRE | 0.31 [0.26 to 0.36] | 0.33 [0.27 to 0.40] | 0.24 [0.19 to 0.30]
  Anti-1, M2: number analyzed (Participants) | 0 | 79 | 76
  Anti-1, M2 |  | 4.19 [3.31 to 5.31] | 2.32 [1.88 to 2.87]
  Anti-4, PRE: number analyzed (Participants) | 165 | 76 | 75
  Anti-4, PRE | 0.45 [0.38 to 0.53] | 0.57 [0.45 to 0.72] | 0.49 [0.39 to 0.61]
  Anti-4, M2: number analyzed (Participants) | 0 | 81 | 77
  Anti-4, M2 |  | 7.80 [6.32 to 9.61] | 4.05 [3.30 to 4.97]
  Anti-5, PRE: number analyzed (Participants) | 166 | 78 | 78
  Anti-5, PRE | 0.61 [0.53 to 0.71] | 0.55 [0.45 to 0.67] | 0.48 [0.39 to 0.59]
  Anti-5, M2: number analyzed (Participants) | 0 | 81 | 77
  Anti-5, M2 |  | 4.65 [3.86 to 5.62] | 3.22 [2.75 to 3.78]
  Anti-6B, PRE: number analyzed (Participants) | 163 | 75 | 76
  Anti-6B, PRE | 0.57 [0.46 to 0.70] | 0.53 [0.40 to 0.69] | 0.48 [0.36 to 0.64]
  Anti-6B, M2: number analyzed (Participants) | 0 | 78 | 76
  Anti-6B, M2 |  | 2.95 [2.23 to 3.91] | 2.18 [1.77 to 2.69]
  Anti-7F, PRE: number analyzed (Participants) | 161 | 73 | 75
  Anti-7F, PRE | 0.79 [0.69 to 0.90] | 0.95 [0.80 to 1.14] | 0.71 [0.58 to 0.87]
  Anti-7F, M2: number analyzed (Participants) | 0 | 81 | 77
  Anti-7F, M2 |  | 6.49 [5.50 to 7.65] | 3.85 [3.18 to 4.66]
  Anti-9V, PRE: number analyzed (Participants) | 164 | 76 | 75
  Anti-9V, PRE | 0.79 [0.67 to 0.92] | 0.85 [0.68 to 1.06] | 0.75 [0.61 to 0.93]
  Anti-9V, M2: number analyzed (Participants) | 0 | 81 | 77
  Anti-9V, M2 |  | 5.31 [4.28 to 6.59] | 3.07 [2.53 to 3.73]
  Anti-14, PRE: number analyzed (Participants) | 168 | 78 | 76
  Anti-14, PRE | 1.30 [1.09 to 1.56] | 1.37 [1.06 to 1.77] | 1.29 [0.97 to 1.72]
  Anti-14, M2: number analyzed (Participants) | 0 | 81 | 77
  Anti-14, M2 |  | 10.60 [8.63 to 13.01] | 6.79 [5.51 to 8.36]
  Anti-18C, PRE: number analyzed (Participants) | 168 | 78 | 78
  Anti-18C, PRE | 0.79 [0.67 to 0.94] | 0.82 [0.61 to 1.10] | 0.87 [0.68 to 1.11]
  Anti-18C, M2: number analyzed (Participants) | 0 | 80 | 77
  Anti-18C, M2 |  | 7.78 [6.21 to 9.74] | 14.14 [11.08 to 18.04]
  Anti-19F, PRE: number analyzed (Participants) | 166 | 75 | 76
  Anti-19F, PRE | 1.36 [1.10 to 1.68] | 1.35 [0.97 to 1.88] | 1.08 [0.78 to 1.50]
  Anti-19F, M2: number analyzed (Participants) | 0 | 78 | 77
  Anti-19F, M2 |  | 16.90 [13.83 to 20.65] | 12.35 [10.23 to 14.91]
  Anti-23F, PRE: number analyzed (Participants) | 165 | 77 | 77
  Anti-23F, PRE | 0.62 [0.51 to 0.76] | 0.67 [0.48 to 0.92] | 0.53 [0.39 to 0.70]
  Anti-23F, M2: number analyzed (Participants) | 0 | 81 | 77
  Anti-23F, M2 |  | 5.25 [4.06 to 6.79] | 2.72 [2.15 to 3.43]

5. Secondary Outcome: Cross-reactive Anti-pneumococcal Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in µg/mL. The pneumococcal serotypes assessed were 6A and 19A (anti-6A and anti-19A) via the 22F-inhibition ELISA. GMCs post Dose 2 are not presented for Nimenrix + Synflorix Group, as they received only one study vaccination dose.
Time Frame: Before vaccination (PRE), at one month post dose 1 (Month 1) and at one month post dose 2 (Month 2)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 174 | 81 | 81
μg/mL
  Anti-6A, PRE: number analyzed (Participants) | 166 | 76 | 77
  Anti-6A, PRE | 0.25 [0.20 to 0.31] | 0.25 [0.19 to 0.35] | 0.26 [0.20 to 0.35]
  Anti-6A, M1: number analyzed (Participants) | 173 | 75 | 81
  Anti-6A, M1 | 1.54 [1.22 to 1.96] | 0.28 [0.20 to 0.39] | 2.07 [1.56 to 2.76]
  Anti-6A, M2: number analyzed (Participants) | 0 | 81 | 77
  Anti-6A, M2 |  | 1.59 [1.10 to 2.31] | 1.30 [0.98 to 1.71]
  Anti-19A, PRE: number analyzed (Participants) | 166 | 75 | 76
  Anti-19A, PRE | 0.17 [0.14 to 0.21] | 0.18 [0.13 to 0.25] | 0.16 [0.12 to 0.21]
  Anti-19A, M1: number analyzed (Participants) | 174 | 77 | 79
  Anti-19A, M1 | 2.00 [1.58 to 2.52] | 0.22 [0.16 to 0.30] | 2.50 [1.89 to 3.30]
  Anti-19A, M2: number analyzed (Participants) | 0 | 79 | 76
  Anti-19A, M2 |  | 2.21 [1.58 to 3.09] | 1.51 [1.12 to 2.04]

6. Secondary Outcome: Opsonophagocytic Titers Against Pneumococcal Serotypes
Description: Opsonophagocytic titers are presented as geometric mean titers (GMTs). The pneumococcal serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (OPSONO-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F). GMTs post Dose 2 are not presented for Nimenrix + Synflorix Group, as they received only one study vaccination dose.
Time Frame: Before vaccination (PRE), at one month post dose 1 (Month 1) and at one month post dose 2 (Month 2)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 68 | 28 | 27
Titers
  Opsono-1, PRE | 6.6 [5.1 to 8.7] | 5.8 [4.0 to 8.4] | 6.2 [4.0 to 9.9]
  Opsono-1, M1: number analyzed (Participants) | 56 | 20 | 26
  Opsono-1, M1 | 395.3 [244.4 to 639.6] | 8.2 [4.4 to 15.3] | 438.6 [224.4 to 857.2]
  Opsono-1, M2: number analyzed (Participants) | 0 | 15 | 26
  Opsono-1, M2 |  | 200.8 [86.1 to 468.2] | 238.0 [117.5 to 482.0]
  Opsono-4, PRE: number analyzed (Participants) | 54 | 23 | 22
  Opsono-4, PRE | 13.7 [7.6 to 24.5] | 14.9 [6.7 to 32.9] | 24.9 [9.0 to 68.6]
  Opsono-4, M1: number analyzed (Participants) | 58 | 16 | 26
  Opsono-4, M1 | 2638.7 [1938.8 to 3591.1] | 10.3 [5.3 to 19.8] | 3621.3 [2488.8 to 5269.1]
  Opsono-4, M2: number analyzed (Participants) | 0 | 15 | 25
  Opsono-4, M2 |  | 2536.5 [1485.3 to 4331.9] | 1427.7 [683.8 to 2980.6]
  Opsono-5, PRE: number analyzed (Participants) | 67 | 28 | 26
  Opsono-5, PRE | 12.9 [9.6 to 17.3] | 10.8 [7.1 to 16.4] | 12.7 [7.7 to 20.9]
  Opsono-5, M1: number analyzed (Participants) | 59 | 19 | 26
  Opsono-5, M1 | 362.1 [261.6 to 501.2] | 11.0 [5.9 to 20.6] | 332.7 [227.2 to 487.1]
  Opsono-5, M2: number analyzed (Participants) | 0 | 15 | 24
  Opsono-5, M2 |  | 233.3 [132.0 to 412.2] | 308.9 [188.2 to 506.9]
  Opsono-6B, PRE: number analyzed (Participants) | 59 | 23 | 20
  Opsono-6B, PRE | 37.4 [20.4 to 68.5] | 26.1 [11.0 to 61.9] | 42.7 [12.5 to 146.5]
  Opsono-6B, M1: number analyzed (Participants) | 57 | 16 | 23
  Opsono-6B, M1 | 678.9 [422.1 to 1091.9] | 56.1 [16.9 to 186.8] | 1158.7 [539.3 to 2489.4]
  Opsono-6B, M2: number analyzed (Participants) | 0 | 15 | 25
  Opsono-6B, M2 |  | 1112.1 [402.1 to 3075.8] | 560.6 [223.6 to 1405.3]
  Opsono-7F, PRE: number analyzed (Participants) | 62 | 24 | 23
  Opsono-7F, PRE | 1795.6 [1416.5 to 2276.1] | 1588.3 [1103.6 to 2286.0] | 1843.1 [1385.7 to 2451.6]
  Opsono-7F, M1: number analyzed (Participants) | 55 | 18 | 23
  Opsono-7F, M1 | 5485.4 [4608.2 to 6529.5] | 2051.2 [1304.0 to 3226.5] | 5421.5 [3948.8 to 7443.5]
  Opsono-7F, M2: number analyzed (Participants) | 0 | 15 | 22
  Opsono-7F, M2 |  | 5235.8 [2619.9 to 10463.7] | 4444.3 [2918.5 to 6768.0]
  Opsono-9V, PRE: number analyzed (Participants) | 60 | 25 | 24
  Opsono-9V, PRE | 728.3 [553.7 to 957.9] | 627.7 [427.3 to 921.9] | 1269.8 [798.4 to 2019.4]
  Opsono-9V, M1: number analyzed (Participants) | 57 | 20 | 24
  Opsono-9V, M1 | 2697.7 [2191.1 to 3321.4] | 445.2 [218.9 to 905.5] | 4862.0 [3345.5 to 7065.9]
  Opsono-9V, M2: number analyzed (Participants) | 0 | 15 | 24
  Opsono-9V, M2 |  | 2709.7 [1635.5 to 4489.5] | 3392.6 [2236.5 to 5146.4]
  Opsono-14, PRE: number analyzed (Participants) | 59 | 25 | 22
  Opsono-14, PRE | 329.5 [228.7 to 474.9] | 324.7 [161.5 to 652.9] | 320.5 [155.6 to 660.3]
  Opsono-14, M1: number analyzed (Participants) | 58 | 18 | 26
  Opsono-14, M1 | 3178.4 [2423.1 to 4169.1] | 214.3 [69.3 to 663.1] | 3914.0 [2506.7 to 6111.5]
  Opsono-14, M2: number analyzed (Participants) | 0 | 15 | 24
  Opsono-14, M2 |  | 2563.7 [1531.3 to 4292.1] | 2149.0 [1381.5 to 3342.8]
  Opsono-18C, PRE: number analyzed (Participants) | 58 | 22 | 26
  Opsono-18C, PRE | 13.9 [8.1 to 24.0] | 10.5 [5.1 to 21.6] | 13.2 [6.6 to 26.2]
  Opsono-18C, M1: number analyzed (Participants) | 55 | 17 | 23
  Opsono-18C, M1 | 1969.9 [1340.0 to 2895.9] | 8.2 [3.7 to 18.2] | 5616.8 [3209.6 to 9829.3]
  Opsono-18C, M2: number analyzed (Participants) | 0 | 15 | 22
  Opsono-18C, M2 |  | 1229.9 [668.5 to 2263.0] | 4190.1 [2326.8 to 7545.6]
  Opsono-19F, PRE: number analyzed (Participants) | 67 | 28 | 27
  Opsono-19F, PRE | 33.5 [21.2 to 52.9] | 34.2 [15.5 to 75.1] | 32.9 [14.7 to 73.4]
  Opsono-19F, M1: number analyzed (Participants) | 57 | 19 | 24
  Opsono-19F, M1 | 2074.7 [1456.3 to 2955.6] | 57.3 [19.0 to 172.5] | 2534.2 [1794.5 to 3578.8]
  Opsono-19F, M2: number analyzed (Participants) | 0 | 15 | 22
  Opsono-19F, M2 |  | 2110.4 [1192.5 to 3734.8] | 1260.4 [788.8 to 2013.8]
  Opsono-23F, PRE: number analyzed (Participants) | 60 | 23 | 23
  Opsono-23F, PRE | 262.3 [128.9 to 533.7] | 98.1 [27.6 to 348.2] | 460.2 [139.7 to 1515.3]
  Opsono-23F, M1: number analyzed (Participants) | 58 | 15 | 26
  Opsono-23F, M1 | 3808.8 [2708.9 to 5355.4] | 199.0 [33.9 to 1168.7] | 3794.6 [2392.0 to 6019.9]
  Opsono-23F, M2: number analyzed (Participants) | 0 | 15 | 26
  Opsono-23F, M2 |  | 3432.4 [2187.3 to 5386.3] | 3284.2 [2184.6 to 4937.3]

7. Secondary Outcome: Opsonophagocytic Titers Against Cross-reactive Pneumococcal Serotypes
Description: Opsonophagocytic titers are presented as geometric mean titers (GMTs). The pneumococcal serotypes assessed were 6A and 19A (OPSONO-6A and OPSONO-19A). GMTs post Dose 2 are not presented for Nimenrix + Synflorix Group, as they received only one study vaccination dose.
Time Frame: Before vaccination (PRE), at one month post dose 1 (Month 1) and at one month post dose 2 (Month 2)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 68 | 27 | 27
Titers
  OPSONO-6A, PRE: number analyzed (Participants) | 58 | 26 | 19
  OPSONO-6A, PRE | 55.8 [30.1 to 103.5] | 73.1 [30.6 to 174.7] | 127.6 [48.9 to 333.0]
  OPSONO-6A, M1: number analyzed (Participants) | 51 | 16 | 22
  OPSONO-6A, M1 | 355.2 [188.7 to 668.8] | 59.4 [17.4 to 202.7] | 696.6 [359.9 to 1348.2]
  OPSONO-6A, M2: number analyzed (Participants) | 0 | 15 | 19
  OPSONO-6A, M2 |  | 566.0 [210.4 to 1522.8] | 284.1 [105.4 to 765.5]
  OPSONO-19A, PRE | 5.3 [4.1 to 6.9] | 5.9 [3.6 to 9.6] | 7.0 [3.8 to 13.2]
  OPSONO-19A, M1: number analyzed (Participants) | 57 | 20 | 24
  OPSONO-19A, M1 | 100.2 [50.3 to 199.5] | 6.3 [3.5 to 11.3] | 214.5 [75.3 to 611.0]
  OPSONO-19A, M2: number analyzed (Participants) | 0 | 15 | 23
  OPSONO-19A, M2 |  | 203.2 [57.6 to 716.6] | 86.8 [28.2 to 267.2]

8. Secondary Outcome: Anti-protein D (Anti-PD) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per milliliter (EL.U/mL). GMCs post Dose 2 are not presented for Nimenrix + Synflorix Group, as they received only one study vaccination dose.
Time Frame: Before vaccination (PRE), at one month post dose 1(Month 1) and at one month post dose 2 (Month 2)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 81 | 43 | 40
EL.U/mL
  Anti-PD, PRE: number analyzed (Participants) | 72 | 37 | 35
  Anti-PD, PRE | 588.4 [455.9 to 759.4] | 633.4 [444.0 to 903.4] | 514.6 [352.1 to 752.1]
  Anti-PD, M1 | 2340.3 [1882.6 to 2909.3] | 632.6 [468.1 to 854.9] | 2452.3 [1790.1 to 3359.6]
  Anti-PD, M2: number analyzed (Participants) | 0 | 43 | 38
  Anti-PD, M2 |  | 2921.6 [2053.6 to 4156.4] | 1854.3 [1313.1 to 2618.4]

9. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW -135 and rSBA-Men-Y Antibody Titers
Description: Antibody titers are presented as geometric mean titers (GMTs) and measured in titers. GMTs post Dose 2 are not presented for Nimenrix + Synflorix Group, as they received only one study vaccination dose.
Time Frame: Before vaccination (PRE) and at one month post dose 2 (Month 2)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 172 | 81 | 79
Titers
  rSBA-MenA, PRE: number analyzed (Participants) | 148 | 69 | 69
  rSBA-MenA, PRE | 15.2 [10.8 to 21.4] | 15.3 [9.3 to 25.2] | 39.4 [22.1 to 70.5]
  rSBA-MenA, M2: number analyzed (Participants) | 0 | 80 | 78
  rSBA-MenA, M2 |  | 4746.8 [3568.4 to 6314.3] | 5288.0 [4498.0 to 6216.9]
  rSBA-MenC, PRE: number analyzed (Participants) | 172 | 81 | 78
  rSBA-MenC, PRE | 5.8 [4.9 to 6.9] | 6.1 [4.7 to 8.0] | 7.7 [5.6 to 10.7]
  rSBA-MenC, M2: number analyzed (Participants) | 0 | 81 | 78
  rSBA-MenC, M2 |  | 1834.6 [1408.1 to 2390.4] | 1579.9 [1218.9 to 2048.0]
  rSBA-MenW, PRE: number analyzed (Participants) | 165 | 75 | 73
  rSBA-MenW, PRE | 46.4 [33.7 to 63.7] | 32.7 [19.8 to 53.9] | 39.6 [23.9 to 65.4]
  rSBA-MenW, M2: number analyzed (Participants) | 0 | 81 | 78
  rSBA-MenW, M2 |  | 5817.6 [4390.8 to 7708.0] | 7666.8 [6502.8 to 9039.0]
  rSBA-MenY, PRE: number analyzed (Participants) | 171 | 78 | 79
  rSBA-MenY, PRE | 66.0 [46.6 to 93.6] | 74.4 [44.7 to 123.9] | 77.0 [45.5 to 130.4]
  rSBA-MenY, M2: number analyzed (Participants) | 0 | 81 | 78
  rSBA-MenY, M2 |  | 4669.5 [3735.6 to 5836.8] | 6461.1 [5329.3 to 7833.2]

10. Secondary Outcome: Anti-meningococcal Polysaccharide (Anti-PS) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in micrograms per milliliter (µg/mL). GMCs post Dose 2 are not presented for Nimenrix + Synflorix Group, as they received only one study vaccination dose.
Time Frame: Before vaccination (PRE), at one month post dose 1 (Month 1) and at one month post dose 2 (Month 2)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 78 | 43 | 40
μg/mL
  Anti-PSA, PRE: number analyzed (Participants) | 73 | 42 | 39
  Anti-PSA, PRE | 0.18 [0.16 to 0.21] | 0.17 [0.15 to 0.19] | 0.20 [0.16 to 0.25]
  Anti-PSA, M1: number analyzed (Participants) | 72 | 36 | 34
  Anti-PSA, M1 | 56.44 [44.38 to 71.77] | 41.94 [26.38 to 66.67] | 0.19 [0.15 to 0.23]
  Anti-PSA, M2: number analyzed (Participants) | 0 | 40 | 35
  Anti-PSA, M2 |  | 18.88 [12.55 to 28.41] | 19.80 [14.68 to 26.71]
  Anti-PSC, PRE: number analyzed (Participants) | 77 | 42 | 40
  Anti-PSC, PRE | 0.16 [0.15 to 0.17] | 0.15 [0.15 to 0.15] | 0.16 [0.15 to 0.17]
  Anti-PSC, M1: number analyzed (Participants) | 78 | 39 | 37
  Anti-PSC, M1 | 24.11 [19.41 to 29.95] | 24.54 [17.77 to 33.89] | 0.16 [0.14 to 0.17]
  Anti-PSC, M2: number analyzed (Participants) | 0 | 43 | 36
  Anti-PSC, M2 |  | 11.56 [8.62 to 15.51] | 9.62 [7.33 to 12.63]
  Anti-PSW-135, PRE: number analyzed (Participants) | 71 | 38 | 35
  Anti-PSW-135, PRE | 0.15 [0.15 to 0.16] | 0.16 [0.14 to 0.19] | 0.15 [0.15 to 0.15]
  Anti-PSW-135, M1: number analyzed (Participants) | 78 | 39 | 36
  Anti-PSW-135, M1 | 12.11 [9.52 to 15.41] | 11.68 [8.06 to 16.92] | 0.15 [0.15 to 0.15]
  Anti-PSW-135, M2: number analyzed (Participants) | 0 | 42 | 35
  Anti-PSW-135, M2 |  | 11.38 [8.10 to 15.98] | 6.75 [4.94 to 9.22]
  Anti-PSY, PRE: number analyzed (Participants) | 74 | 40 | 37
  Anti-PSY, PRE | 0.15 [0.15 to 0.15] | 0.17 [0.14 to 0.19] | 0.16 [0.14 to 0.17]
  Anti-PSY, M1: number analyzed (Participants) | 77 | 38 | 37
  Anti-PSY, M1 | 12.03 [9.63 to 15.02] | 10.78 [7.24 to 16.05] | 0.15 [0.15 to 0.16]
  Anti-PSY, M2: number analyzed (Participants) | 0 | 42 | 35
  Anti-PSY, M2 |  | 10.22 [7.24 to 14.41] | 8.47 [6.45 to 11.10]

11. Secondary Outcome: Anti-tetanus (Anti-T) Antibody Concentrations
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in international units per milliliter (IU/mL). GMCs post Dose 2 are not presented for Nimenrix + Synflorix Group, as they received only one study vaccination dose.
Time Frame: Before vaccination (PRE), at one month post dose 1 (Month 1) and at one month post dose 2 (Month 2)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 79 | 42 | 39
IU/mL
  Anti-T, PRE: number analyzed (Participants) | 79 | 42 | 38
  Anti-T, PRE | 0.499 [0.399 to 0.624] | 0.566 [0.428 to 0.749] | 0.502 [0.385 to 0.654]
  Anti-T, M1: number analyzed (Participants) | 78 | 39 | 39
  Anti-T, M1 | 18.446 [14.797 to 22.995] | 18.137 [12.085 to 27.218] | 4.412 [3.298 to 5.901]
  Anti-T, M2: number analyzed (Participants) | 0 | 42 | 37
  Anti-T, M2 |  | 16.643 [12.460 to 22.230] | 13.773 [10.932 to 17.352]

12. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site.
Time Frame: Within the 4-day (Days 0-3) post-vaccination period after each dose
Population: The analysis was done on the Total Vaccinated cohort, which included all vaccinated subjects with the symptoms sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 180 | 91 | 88
Participants
  Any Pain, Dose 1, Synflorix: number analyzed (Participants) | 180 | 0 | 88
  Any Pain, Dose 1, Synflorix | 90 | 0 | 47
  Grade 3 Pain, Dose 1, Synflorix: number analyzed (Participants) | 180 | 0 | 88
  Grade 3 Pain, Dose 1, Synflorix | 14 | 0 | 6
  Any Pain, Dose 1, Nimenrix: number analyzed (Participants) | 180 | 91 | 0
  Any Pain, Dose 1, Nimenrix | 87 | 40 | 0
  Grade 3 Pain, Dose 1, Nimenrix: number analyzed (Participants) | 180 | 91 | 0
  Grade 3 Pain, Dose 1, Nimenrix | 14 | 4 | 0
  Any Redness, Dose 1, Synflorix: number analyzed (Participants) | 180 | 0 | 88
  Any Redness, Dose 1, Synflorix | 54 | 0 | 32
  Grade 3 Redness, Dose 1, Synflorix: number analyzed (Participants) | 180 | 0 | 88
  Grade 3 Redness, Dose 1, Synflorix | 2 | 0 | 4
  Any Redness, Dose 1, Nimenrix: number analyzed (Participants) | 180 | 91 | 0
  Any Redness, Dose 1, Nimenrix | 56 | 31 | 0
  Grade 3 Redness, Dose 1, Nimenrix: number analyzed (Participants) | 180 | 91 | 0
  Grade 3 Redness, Dose 1, Nimenrix | 3 | 1 | 0
  Any Swelling, Dose 1, Synflorix: number analyzed (Participants) | 180 | 0 | 88
  Any Swelling, Dose 1, Synflorix | 70 | 0 | 42
  Grade 3 Swelling, Dose 1, Synflorix: number analyzed (Participants) | 180 | 0 | 88
  Grade 3 Swelling, Dose 1, Synflorix | 3 | 0 | 3
  Any Swelling, Dose 1, Nimenrix: number analyzed (Participants) | 180 | 91 | 0
  Any Swelling, Dose 1, Nimenrix | 66 | 37 | 0
  Grade 3 Swelling, Dose 1, Nimenrix: number analyzed (Participants) | 180 | 91 | 0
  Grade 3 Swelling, Dose 1, Nimenrix | 3 | 1 | 0
  Any Pain, Dose 2, Synflorix: number analyzed (Participants) | 0 | 91 | 0
  Any Pain, Dose 2, Synflorix | 0 | 43 | 0
  Grade 3 Pain, Dose 2, Synflorix: number analyzed (Participants) | 0 | 91 | 0
  Grade 3 Pain, Dose 2, Synflorix | 0 | 8 | 0
  Any Pain, Dose 2, Nimenrix: number analyzed (Participants) | 0 | 0 | 85
  Any Pain, Dose 2, Nimenrix | 0 | 0 | 34
  Grade 3, Dose 2, Nimenrix: number analyzed (Participants) | 0 | 0 | 85
  Grade 3, Dose 2, Nimenrix | 0 | 0 | 2
  Any Redness, Dose 2, Synflorix: number analyzed (Participants) | 0 | 91 | 0
  Any Redness, Dose 2, Synflorix | 0 | 29 | 0
  Grade 3 Redness, Dose 2, Synflorix: number analyzed (Participants) | 0 | 91 | 0
  Grade 3 Redness, Dose 2, Synflorix | 0 | 3 | 0
  Any Redness, Dose 2, Nimenrix: number analyzed (Participants) | 0 | 0 | 85
  Any Redness, Dose 2, Nimenrix | 0 | 0 | 24
  Grade 3 Redness, Dose 2, Nimenrix: number analyzed (Participants) | 0 | 0 | 85
  Grade 3 Redness, Dose 2, Nimenrix | 0 | 0 | 1
  Any Swelling, Dose 2, Synflorix: number analyzed (Participants) | 0 | 91 | 0
  Any Swelling, Dose 2, Synflorix | 0 | 38 | 0
  Grade 3 Swelling, Dose 2, Synflorix: number analyzed (Participants) | 0 | 91 | 0
  Grade 3 Swelling, Dose 2, Synflorix | 0 | 1 | 0
  Any Swelling, Dose 2, Nimenrix: number analyzed (Participants) | 0 | 0 | 85
  Any Swelling, Dose 2, Nimenrix | 0 | 0 | 30
  Grade 3 Swelling, Dose 2, Nimenrix: number analyzed (Participants) | 0 | 0 | 85
  Grade 3 Swelling, Dose 2, Nimenrix | 0 | 0 | 2

13. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and temperature [defined as rectally temperature equal to or above (≥) 38.0 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 drowsiness = drowsiness that prevented normal activities. Grade 3 irritability = crying that could not be comforted/ prevented normal activity. Grade 3 loss of appetite = not eating at all. Grade 3 fever = fever higher than (>) 40.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within the 4-day (Days 0-3) post-vaccination period after each dose
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 180 | 91 | 88
Participants
  Any Drowsiness, Dose 1 | 59 | 21 | 35
  Grade 3 Drowsiness, Dose 1 | 1 | 0 | 1
  Related Drowsiness, Dose 1 | 55 | 18 | 34
  Any Irritability, Dose 1 | 72 | 33 | 43
  Grade 3 Irritability, Dose 1 | 2 | 0 | 1
  Related Irritability, Dose 1 | 65 | 30 | 40
  Any Loss of appetite, Dose 1 | 55 | 22 | 33
  Grade 3 Loss of appetite, Dose 1 | 2 | 0 | 1
  Related Loss of appetite, Dose 1 | 46 | 18 | 28
  Any Temperature, Dose 1 | 25 | 10 | 15
  Grade 3 Temperature, Dose 1 | 0 | 0 | 0
  Related Temperature, Dose 1 | 24 | 10 | 15
  Any Drowsiness, Dose 2: number analyzed (Participants) | 0 | 91 | 85
  Any Drowsiness, Dose 2 | 0 | 25 | 17
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 0 | 91 | 85
  Grade 3 Drowsiness, Dose 2 | 0 | 1 | 0
  Related Drowsiness, Dose 2: number analyzed (Participants) | 0 | 91 | 85
  Related Drowsiness, Dose 2 | 0 | 22 | 15
  Any Irritability, Dose 2: number analyzed (Participants) | 0 | 91 | 85
  Any Irritability, Dose 2 | 0 | 35 | 29
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 0 | 91 | 85
  Grade 3 Irritability, Dose 2 | 0 | 1 | 1
  Related Irritability, Dose 2: number analyzed (Participants) | 0 | 91 | 85
  Related Irritability, Dose 2 | 0 | 30 | 25
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 0 | 91 | 85
  Any Loss of appetite, Dose 2 | 0 | 22 | 22
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 0 | 91 | 85
  Grade 3 Loss of appetite, Dose 2 | 0 | 0 | 0
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 0 | 91 | 85
  Related Loss of appetite, Dose 2 | 0 | 20 | 20
  Any Temperature, Dose 2: number analyzed (Participants) | 0 | 91 | 85
  Any Temperature, Dose 2 | 0 | 18 | 11
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 0 | 91 | 85
  Grade 3 Temperature, Dose 2 | 0 | 1 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 0 | 91 | 85
  Related Temperature, Dose 2 | 0 | 16 | 9

14. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within the 31-day (Day 0-30) post-vaccination period after each dose
Population: The analysis was done on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 182 | 91 | 90
Participants
  Any AE(s) post-Dose 1 | 82 | 39 | 42
  Any AE(s) post-Dose 2 | 0 | 40 | 31

15. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Throughout the entire study duration (Day 0-Month 7)
Population: The analysis was done on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 182 | 91 | 90
Participants | 6 | 3 | 4

16. Secondary Outcome: Number of Subjects Reporting Rash
Description: Rash-like symptoms assessed were hives, idiopathic thrombocytopenic purpura, petechiae.
Time Frame: Throughout the entire study duration (Day 0-Month 7)
Population: The analysis was done on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 182 | 91 | 90
Participants | 9 | 10 | 5

17. Secondary Outcome: Number of Subjects With New Onset Chronic Illnesses (NOCIs)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: Throughout the entire study duration (Day 0-Month 7)
Population: The analysis was done on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 182 | 91 | 90
Participants | 0 | 1 | 0

18. Secondary Outcome: Number of Subjects Reporting Adverse Events Resulting in Emergency Room (ER) Visits
Description: Among AEs prompting emergency room visits were: infections, injuries, skin diseases, gastrointestinal symptoms.
Time Frame: Throughout the entire study duration (Day 0-Month 7)
Population: The analysis was done on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
Number analyzed (Participants) | 182 | 91 | 90
Participants | 13 | 10 | 9

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 4-day post-vaccination period (Days 0-3). Unsolicited AEs: during the 31-day post-vaccination period (Days 0-30). SAEs: during the entire study period (from Day 0 up to Month 7).
Arm/Group | Nimenrix + Synflorix Group | Nimenrix Group | Synflorix Group
All-Cause Mortality (participants affected / at risk) | 0/182 | 0/91 | 0/90
Serious Adverse Events (participants affected / at risk) | 6/182 | 3/91 | 4/90
Other Adverse Events (participants affected / at risk) | 154/182 | 81/91 | 76/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix + Synflorix Group (N=182) | Nimenrix Group (N=91) | Synflorix Group (N=90)
Bronchopneumonia (Infections and infestations) | 1 | 2 | 0
Croup infectious (Infections and infestations) | 2 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 2
Bronchiolitis (Infections and infestations) | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis bacterial (Infections and infestations) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Infantile asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nimenrix + Synflorix Group (N=182) | Nimenrix Group (N=91) | Synflorix Group (N=90)
Nasopharyngitis (post-Dose 1) (Infections and infestations) | 25 | 15 | 18
Upper respiratory tract infection (post-Dose 1) (Infections and infestations) | 22 | 6 | 9
Nasopharyngitis (post-Dose 2) (Infections and infestations) | 0/0 | 14 | 7
Upper respiratory tract infection (post-Dose 2) (Infections and infestations) | 0/0 | 6 | 5
Upper respiratory tract infection bacterial (post-Dose 2) (Infections and infestations) | 0/0 | 2 | 5
Pain (post-Dose 1 of Synflorix) (General disorders) | 90/180 | 0/0 | 47/88
Pain (post-Dose 1 of Nimenrix) (General disorders) | 87/180 | 40 | 0/0
Redness (post-Dose 1 of Synflorix) (General disorders) | 54/180 | 0/0 | 32/88
Redness (post-Dose 1 of Nimenrix) (General disorders) | 56/180 | 31 | 0/0
Swelling (post-Dose 1 of Synflorix) (General disorders) | 70/180 | 0/0 | 42/88
Swelling (post-Dose 1 of Nimenrix) (General disorders) | 66/180 | 37 | 0/0
Pain (post-Dose 2 of Synflorix) (General disorders) | 0/0 | 43 | 0/0
Pain (post-Dose 2 of Nimenrix) (General disorders) | 0/0 | 0/0 | 34/85
Redness (post-Dose 2 of Synflorix) (General disorders) | 0/0 | 29 | 0/0
Redness (post-Dose 2 of Nimenrix) (General disorders) | 0/0 | 0/0 | 24/85
Swelling (post-Dose 2 of Synflorix) (General disorders) | 0/0 | 38 | 0/0
Swelling (post-Dose 2 of Nimenrix) (General disorders) | 0/0 | 0/0 | 30/85
Drowsiness (post-Dose 1) (General disorders) | 59/180 | 21 | 35/88
Irritability (post-Dose 1) (General disorders) | 72/180 | 33 | 43/88
Loss of appetite (post-Dose 1) (General disorders) | 55/180 | 22 | 33/88
Temperature (post-Dose 1) (General disorders) | 25/180 | 10 | 15/88
Drowsiness (post-Dose 2) (General disorders) | 0/0 | 25 | 17/85
Irritability(post-Dose 2) (General disorders) | 0/0 | 35 | 29/85
Loss of appetite (post-Dose 2) (General disorders) | 0/0 | 22 | 22/85
Temperature (post-Dose 2) (General disorders) | 0/0 | 18 | 11/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.